CLINICAL TRIAL: NCT01606098
Title: The Role of Surgery of the Primary Tumour With Few or Absent Symptoms in Patients With Synchronous Unresectable Metastases of Colorectal Cancer, a Randomized Phase III Study. A Study of the Dutch Colorectal Cancer Group (DCCG)
Brief Title: The Role of Surgery of the Primary Tumour in Patients With Synchronous Unresectable Metastases of Colorectal Cancer
Acronym: CAIRO4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dutch Colorectal Cancer Group (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIRO4
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Colon Cancer; Primary Tumour; Rectal Cancer
Keywords: Surgery; Chemotherapy
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Neoadjuvant Therapy; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Systemic treatment (Active Comparator): First-line fluoropyrimidine-based chemotherapy with bevacizumab initiated within 4 weeks of randomization, followed by salvage therapy upon progression at the discretion of the local investigator. Surgery of primary tumour will be performed only when indicated by local signs or symptoms.
  Interventions: Drug: Systemic treatment
- Surgery followed by systemic treatment (Experimental): Surgery within 4 weeks of randomization followed by fluoropyrimidine-based chemotherapy with bevacizumab until progression or unacceptable toxicity, followed by salvage therapy upon progression at the discretion of the local investigator
  Interventions: Procedure: Surgery of the primary tumour; Drug: Systemic treatment

INTERVENTIONS:
Procedure: Surgery of the primary tumour — Surgical resection of the colon tumour
  Arms: Surgery followed by systemic treatment
Drug: Systemic treatment — First line fluoropyrimidine-based chemotherapy with bevacizumab. The chemotherapy regimen is to the discretion of the local investigator, who may choose between:
  5FU/LV or capecitabine or capecitabine + oxaliplatin(CAPOX)or 5FU + oxaliplatin(FOLFOX 4 or FOLFOX 7)or 5FU + irinotecan (FOLFIRI) or capecitabine + irinotecan(CAPIRI)
  Other Names: Bevacizumab in combination with fluoropyrimidine-based schedules

SUMMARY:
The clinical benefit of resection of the primary tumour in patients with synchronous unresectable metastases is not known. In the literature studies usually describe retrospective selected patients with synchronous metastases treated with or without resection of the primary tumour. All these studies are biased in patient selection and there are no prospective randomized studies on this topic. In patients with few or absent symptoms of the primary tumour, arguments both in favour and against initial resection have been presented, and therefore a randomized trial is warranted. Although recent publications suggest that resection of the primary tumour in synchronous metastasized colon cancer patients might not be necessary, this appears to be based on feasibility and not on clinical outcome. Several studies comparing large groups of patients with or without resection of the primary tumour suggest an improved survival when the primary tumour is resected. A potential benefit of resection of the primary tumour is to prevent complications of the primary tumour during chemotherapy treatment or during later stages of the disease. A recent analysis of the CAIRO and CAIRO2 data showed that metastatic colon cancer patients who had a resection of the primary tumour prior to study entry, had an improved survival compared to patients without a resection of the primary tumour. However, these patients were selected after the primary tumour was resected and therefore these results are not corrected for surgical morbidity and mortality. The investigators here propose a randomized trial in order to demonstrate that resection of the primary tumour does improve overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of colorectal cancer
* Resectable primary tumour in situ with unresectable distant metastases
* No indication for neo-adjuvant (chemo)radiation
* No severe signs or symptoms related to the primary tumour (i.e. severe bleeding, obstruction, severe abdominal pain) that require immediate surgery or other symptomatic treatment (e.g. stenting)
* No prior systemic treatment for advanced disease
* Age ≥ 18 years
* WHO performance status 0-2
* Laboratory values obtained ≤ 4 weeks prior to randomization: Adequate bone marrow function (Hb ≥ 6.0 mmol/L, absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L), renal function (serum creatinine ≤ 1.5x ULN and creatinine clearance, Cockroft formula, ≥ 30 ml/min), liver function (serum bilirubin ≤ 2 x ULN, serum transaminases ≤ 3 x ULN without presence of liver metastases or ≤ 5x ULN with presence of liver metastases)
* Expected adequacy of follow-up
* Written informed consent
* CT scan abdomen and CT thorax/X-thorax performed ≤ 4 weeks prior to randomization

Exclusion Criteria:

* Pregnancy, lactation
* Unresectable primary tumour (i.e. neurovascular encasement, substantial ingrowth in pancreatic head), or any condition preventing the safety or feasibility of resection of the primary tumour, i.e. massive ascites or extensive peritoneal disease
* Requirement of neoadjuvant (chmo)radiation therapy
* Second primary malignancy within the past 5 years with the exception of adequately treated in situ carcinoma of any organ or basal cell carcinoma of the skin
* Any medical condition that prevents the safe administration of systemic treatment
* Previous intolerance of fluoropyrimidines, known dihydropyrimidine dehydrogenase (DPD) deficiency
* Planned radical resection of all metastatic disease
* Uncontrolled hypertension, i.e. values consistently > 150/100 mmHg
* Use of ≥ 3 antihypertensive drugs
* Significant cardiovascular disease < 1 yr before randomization (symptomatic congestive heart failure, myocardial infarction, unstable angina pectoris, serious uncontrolled cardiac arrhythmia, cerebro vascular event)
* Chronic active infection
* Concurrent treatment with any other anti-cancer therapy as described per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | Time from randomisation until death, assessed up to 5 years
  Overall survival of the intent-to-treat population

SECONDARY OUTCOMES:
Progression-free survival | Time from randomisation until first progression or death whichever comes first, asessed up to 5 years
Response to chemotherapy | Fist-line chemotherapy, assessed until progression
  Response rate according to RECIST 1.1
Systemic therapy related toxicity | Every 3 weeks during first-line treatment
  Adverse events grade 3-4 according to NCI-CTC 4.0
Surgery related morbidity and mortality | 30 days
Quality of life | Every 6 months from randomisation until first progression
  EORTC QLQ-C30 and CR38
Interval between randomization and initiation of systemic treatment | Number of days between randomization and initiation of systemic treatment
Cost-benefit analyses | Until end of first-line systemic treatment
Patients requiring resection of the primary tumour in the non-resection arm | Time from randomisation until death, assessed up to 5 years
  Number of patients requiring resection of the primary tumour in the non-resection arm
Overall survival in patients in whom treatment according to protocol was initiated | Time form randomisation until death, assessed up to 5 years
  Having received at least one cycle of systemic treatment in arm A and surgery in arm B

CONTACTS AND LOCATIONS:
Overall Officials: M. Koopman, Prof MD PhD, Principal Investigator — UMC Utrecht; H. JW de Wilt, Prof MD PhD, Principal Investigator — Radboud University Medical Center
Locations (46):
- Denmark (5):
  - University Hospital Aalborg, Aalborg
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Regionshospital Herning, Herning
  - Roskilde hospital, Roskilde
- Netherlands (41):
  - Jeroen Bosch, 's-Hertogenbosch
  - Medisch Centrum Alkmaar, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Flevoziekenhuis, Almere Stad
  - Ziekenhuis Amstelland, Amstelveen
  - Academic Medical Centre, Amsterdam
  - OLVG, Amsterdam
  - VUMC, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Wilhelmina Ziekenhuis, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia Ziekenhuis, Breda
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - St Annaziekenhuis, Geldrop
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - UMCG, Groningen
  - Spaarne Gasthuis, Haarlem
  - St Jansdal, Harderwijk
  - Elkerliek Ziekenhuis, Helmond
  - Spaarne Gasthuis, Hoofddorp
  - St Antonius Ziekenhuis, Nieuwegein
  - Radboudumc, Nijmegen
  - Waterland Ziekenhuis, Purmerend
  - Laurentius Ziekenhuis, Roermond
  - Maasstad Ziekenhuis, Rotterdam
  - Erasmus MC, Rotterdam
  - Fransicus Gastuis & Vlietland, Rotterdam
  - Antonius Ziekenhuis, Sneek
  - MC Haaglanden en Bronovo Nebo, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Elisabeth-Tweesteden, Tilburg
  - Bernhoven Ziekenhuis, Uden
  - University Medical Centre Utrecht, Utrecht
  - Bernhoven Ziekenhuis, Veghel
  - VieCuri Medisch Centrum, Venlo
  - Zaans Medisch Centrum, Zaandam
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Kruijssen DEW, Elias SG, van de Ven PM, van Rooijen KL, Lam-Boer J', Mol L, Punt CJA, Sommeijer DW, Tanis PJ, Nielsen JD, Yilmaz MK, van Riel JMGH, Wasowiz-Kemps DK, Loosveld OJL, van der Schelling GP, de Groot JWB, van Westreenen HL, Jakobsen HL, Fromm AL, Hamberg P, Verseveld M, Jaensch C, Liposits GI, van Duijvendijk P, Oulad Hadj J, van der Hoeven JAB, Trajkovic M, de Wilt JHW, Koopman M; CAIRO4 Working Group. Upfront resection versus no resection of the primary tumor in patients with synchronous metastatic colorectal cancer: the randomized phase III CAIRO4 study conducted by the Dutch Colorectal Cancer Group and the Danish Colorectal Cancer Group. Ann Oncol. 2024 Sep;35(9):769-779. doi: 10.1016/j.annonc.2024.06.001. Epub 2024 Jun 7. PMID 38852675
- [Derived] van der Kruijssen DEW, Elias SG, Vink GR, van Rooijen KL, 't Lam-Boer J, Mol L, Punt CJA, de Wilt JHW, Koopman M; CAIRO4 Working Group. Sixty-Day Mortality of Patients With Metastatic Colorectal Cancer Randomized to Systemic Treatment vs Primary Tumor Resection Followed by Systemic Treatment: The CAIRO4 Phase 3 Randomized Clinical Trial. JAMA Surg. 2021 Dec 1;156(12):1093-1101. doi: 10.1001/jamasurg.2021.4992. PMID 34613339
- [Derived] 't Lam-Boer J, Mol L, Verhoef C, de Haan AF, Yilmaz M, Punt CJ, de Wilt JH, Koopman M. The CAIRO4 study: the role of surgery of the primary tumour with few or absent symptoms in patients with synchronous unresectable metastases of colorectal cancer--a randomized phase III study of the Dutch Colorectal Cancer Group (DCCG). BMC Cancer. 2014 Oct 2;14:741. doi: 10.1186/1471-2407-14-741. PMID 25277170
- See also: Dutch Colorectal Cancer Group — http://www.dccg.nl